CLINICAL TRIAL: NCT06499610
Title: Prospective, Open-label, Single-arm Clinical Study of Irinotecan Liposomes Combined With Cindilizumab and Lunvalatinib as Second-line Treatment for Adenocarcinoma of Advanced Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: Clinical Study of Irinotecan Liposome Combination Therapy for Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Li EnXiao, Doctor Medicinae, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-102
Record Dates: First submitted 2024-07-03; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer
Keywords: Irinotecan lipoposomes; And adenocarcinoma of advanced gastric cancer and gastroesophageal junction; Second line treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): therapeutic measure： Irinotecan hydrochloride for liposome injection 70mg/m2，intravenous drip，d1 Sintilimab Injection 200mg，intravenous drip，d1 Lenvatinib Mesilate Capsules ，8mg (weight<60kg) or 12mg (weight≥60kg) ,po, qd
  Interventions: Drug: Irinotecan Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Irinotecan Hydrochloride Liposome Injection — At the dose of 70mg / m2, for patients homozygous for UGT1A1 * 28, the first dose of irinotecan was adjusted to 50mg / m2,70mg / m2 if the patient tolerated during the first cycle and 70 mg / m 2 in the subsequent cycle; add 500 mL of 5% glucose injection or 0.9% sodium chloride injection for intravenous infusion within 90 minutes. On the first day of each treatment cycle.
  Other Names: Sintilimab Injection; Lenvatinib Mesilate Capsules

SUMMARY:
This study is a single-arm, single-center, exploratory clinical study. It is expected that 44 patients with advanced gastric and gastroesophageal junction adenocarcinoma with first-line treatment failure will be included to receive irinotecan liposomes combined with cindilizumab and renvalatinib. The study unit is the First Affiliated Hospital of Xi'an Jiaotong University. The study included screening period (28 days), treatment period (6 cycles), and follow-up period. Subjects signed the informed consent and underwent baseline examination during the screening period, patients meeting the exclusion criteria entered the treatment period, and all subjects completed the protocol to observe safety, tolerability and efficacy. The same subject received only one dosing schedule during the study period. The follow-up period begins after the end of the treatment period.

DETAILED DESCRIPTION:
This study is an exploratory clinical study. It is expected to include 44 patients with second-line advanced gastric and gastroesophageal junction adenocarcinoma, all treated with irinotecan liposome combined with cindilizumab and lunvatinib.

The dosing regimen of irinotecan liplex injection was 70 mg / m2, cindilizmab 200mg, and valatinib 8-12mg (dose determined by body weight), every 3 weeks, every 2 treatment cycles (every 6 weeks). The subject is scheduled to receive 6 cycles of treatment, or develop intolerable toxicity, or terminate the study for other reasons.

The study included screening period (within 28 days), treatment period (6 cycles) and follow-up period. Subjects signed the informed consent and underwent baseline examination during the screening period, patients meeting the exclusion criteria entered the treatment period, and all subjects completed the protocol to observe safety, tolerability and efficacy. The same subject received only one dosing schedule during the study period. The follow-up period begins after the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* The patient was fully aware of the study and volunteered to participate in and signed the informed consent form (ICF);
* Age≥18 years old;
* Expected survival time of 3 months;
* Patients with pathologically confirmed advanced gastric cancer and adenocarcinoma of the gastroesophageal junction;
* Failure or intolerance of previous first-line anti-tumor therapy;
* CPS 1 was detected by PD-L1 expression level;
* According to RECIST1.1 criteria, the patient has at least one measurable diameter target lesion (long diameter of tumor lesion CT scan 10mm, short diameter of lymph node lesion CT scan 15mm and scanning layer thickness of 5mm);
* Bone marrow function: neutrophils 1.5109 / L, platelets 100109 / L, and hemoglobin 75g / L;
* The ECOG score is 0-2 points;
* Liver and kidney function: upper limit of 1.5 times normal value of serum creatinine; upper limit of normal value of AST and ALT (upper limit of normal value of 5 times for patients with liver invasion); upper limit of normal value of total bilirubin (upper limit of normal value of 3 times for patients with liver invasion);
* Women of childbearing age must have a negative pregnancy test (serum) within 7 days before enrollment, and must be willing to use appropriate methods for contraception during the trial;
* Consent to provide the histological samples;

Exclusion Criteria:

* Allergic reaction to any study drug or its ingredients;
* Patients with severe hepatic and renal insufficiency;
* Have used a strong CYP3A4 inducer within 2 weeks before the first dose of the trial drug, or have used a strong CYP3A4 inhibitor or a strong UGT1A1 inhibitor within 1 week;
* Uncontrollable systemic diseases (such as advanced infection, uncontrolled hypertension, diabetes mellitus, etc.);
* Patients with intestinal obstruction and gastrointestinal bleeding;
* According to the HER 2 testing process and evaluation criteria in CSCO Guidelines for Diagnosis and Treatment of Gastric Cancer 2024 edition: confirmed by immunohistochemistry (IHC), HER2 2 + accompanied by in situ hybridization with gene amplification or HER2 3 +;
* Have any active autoimmune disease or a history of autoimmune disease, such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, and reduced thyroid function (which can be included after normal hormone replacement therapy);
* Heart function and disease are one of the following:

  1. Long QTc syndrome or QTc interval> 480 ms;
  2. Complete left bundle branch block, degree II or III atrioventricular block;
  3. Severe, uncontrolled arrhythmias requiring medical therapy;
  4. New York Society of Cardiology grade III;
  5. Cardiac ejection fraction (LVEF) below 50%;
  6. history of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, clinically severe pericardial disease, or ECG evidence of acute ischemic or active conduction system abnormalities within 6 months prior to recruitment.
* Uncontrolled ascites and abdominal cavity infection;
* Active infection of hepatitis B and C (positive for HBV surface antigen and 1x103 copies / mL and 1x103 copies / mL);
* Human immunodeficiency virus (HIV) infection (HIV antibody positive);
* Previous or current other malignancies (except basal cell carcinoma of the skin with non-melanoma, carcinoma of the breast / cervix in situ, and other malignancies that have been effectively controlled without treatment in the past five years);
* Pregnant and lactating women and patients of childbearing age who are unwilling to take contraception;
* Other investigator judged ineligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression-free survival | Intracranial progression-free survival (PFS) analysis based on investigator assessment and will be assessed up to 3 years.
  Intracranial progression-free survival (PFS) analysis based on investigator assessment and will be assessed up to 3 years.

SECONDARY OUTCOMES:
Intracranial Objective response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The number (%) of patients defined as complete or partial response, assessed using the investigator, version 1.1 (RECIST 1.1), was from the enrollment of subjects to the end of chemotherapy.
Intracranial Disease Control Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The percentage of subjects who have a best response of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by the Investigator, was from the enrollment of subjects to the end of chemotherapy.
Overall Survival | The time from beginning of treatment until death due to any cause and will be assessed up to 3 years.
  Overall survival is defined as the time from beginning of treatment until death due to any cause and will be assessed up to 3 years.
Safety/Adverse event | From the recorded first treatment to 4 weeks after the recorded last treatment
  Incidence of Adverse Events (AEs): Incidence, severity and seriousness of adverse events, incidence of serious adverse events (SAEs), which usually be graded by CTCAE v5.0 based on current clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Enxiao Li, doctor, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China